CLINICAL TRIAL: NCT00497393
Title: Clinical Decision Unit (CDU) - Evaluation of a Novel Approach to Address Emergency Department Overcrowding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Capital Health, Canada (Other)
Responsible Party: Brian Holroyd, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B-130607
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Acute Illness
Keywords: Emergency department, administration, overcrowding
MeSH Terms: conditions — Emergencies; Crowding | interventions — Clinical Observation Units

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Control (No Intervention): regular use of the 2-bed areas in the Emergency department
  Interventions: Behavioral: Clinical Decision Unit

INTERVENTIONS:
Behavioral: Clinical Decision Unit — a dedicated 2-bed area to see patients and then rotate them back into the waiting room area for labs and diagnostic imaging.

SUMMARY:
This randomized controlled trial will introduce a Clinical Decision Unit (CDU) into the University of Alberta Hospital Emergency Department(ED)and assess the influence on ED length of stay, patients who leave without being seen, and other ED Overcrowding outcomes.

DETAILED DESCRIPTION:
The study will take place over a 6-week period that will be spilt into three-two-week blocks. Using computerized blocks of 2 weeks, days of the week will be randomly allocated so that each day of the week receives one intervention (CDU) and one control day for the study period. The CDU involves transforming an ED bed location to a 6-chair internal waiting room with 2 adjacent beds assigned to act as assessment and treatment locations. Patients will transition between the chair and stretcher to optimize the use of ED space.

ELIGIBILITY:
Inclusion Criteria:

* Only adult patients (>17 years of age) presenting to the University of Alberta Hospital Emergency Department (UAH ED), during the study interval will be included in the evaluation.

Exclusion Criteria:

* Direct admits/Pediatric patients.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6217 (Actual)
Dates: Start 2007-07; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Total ED length of stay | in the Emergency Department

SECONDARY OUTCOMES:
Left without being seen (LWBS) rates | in the Emergency Department
nurse and physician satisfaction | following Emergency Department shift
ambulance turnaround times (time | in the Emergency Department

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bullard, MD, Principal Investigator — University of Alberta Hospital, Edmonton, Alberta, T6G 2B7, Canada
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada